CLINICAL TRIAL: NCT00560300
Title: Regulation of Bone Formation in Renal Osteodystrophy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: DK35423 (completed)
Record Dates: First submitted 2007-11-13; First posted 2007-11-19 (Estimated); Last update posted 2010-01-14 (Estimated); Status verified 2010-01

CONDITIONS: Secondary Hyperparathyroidism; Renal Osteodystrophy
MeSH Terms: conditions — Hyperparathyroidism, Secondary; Chronic Kidney Disease-Mineral and Bone Disorder | interventions — 1 alpha-hydroxyergocalciferol; Calcitriol; Sevelamer; Calcium Carbonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): Doxercalciferol + Calcium Carbonate
  Interventions: Drug: 1 alpha D2; Drug: Calcium Carbonate
- 2 (Experimental): Doxercalciferol + Sevelamer
  Interventions: Drug: 1 alpha D2; Drug: Sevelamer HCl
- 3 (Experimental): Calcitriol + Calcium Carbonate
  Interventions: Drug: 1,25 dihydroxy vitamin D3; Drug: Calcium Carbonate
- 4 (Experimental): Calcitriol + Sevelamer
  Interventions: Drug: 1,25 dihydroxy vitamin D3; Drug: Sevelamer HCl

INTERVENTIONS:
Drug: 1 alpha D2 — Vitamin D sterol
  Other Names: Doxercalciferol; Hectoral
  Arms: 1; 2
Drug: 1,25 dihydroxy vitamin D3 — Active vitamin D sterol
  Other Names: Calcitriol; Rocaltrol
  Arms: 3; 4
Drug: Sevelamer HCl — Phosphate binder
  Other Names: Renagel
  Arms: 2; 4
Drug: Calcium Carbonate — Phosphate binder
  Other Names: Tums; Titrilac
  Arms: 1; 3

SUMMARY:
To examine the effects of two types of active vitamin D (calcitriol and doxercalciferol) and two phosphate binders (sevelamer and calcium carbonate) on the bone disease and blood tests of children with kidney failure

DETAILED DESCRIPTION:
Pediatric patients treated with CCPD who displayed biochemical and bone biopsy proven secondary hyperparathyroidism were randomly assigned to one of 2 vitamin D analogues (calcitriol or doxercalciferol) and one of two phosphate binders (sevelamer or calcium carbonate) in a two by two factorial designed prospective trial. Serum biochemical measurements were obtained at baseline and monthly throughout the 8 months of the trial. Bone biopsy was obtaine at baseline and repeated at study completion.

ELIGIBILITY:
Inclusion Criteria:

* Stable end-stage kidney disease treated with continuous cycling peritoneal dialysis,
* Biochemical evidence of secondary hyperparathyroidism (PTH>400 pg/ml) with bone biopsy evidence of high turnover bone disease

Exclusion Criteria:

* History of parathyroidectomy
* Growth hormone
* Prednisone, or other immunosuppressant medication within the past year.
* Recent history of medication non-compliance.

Ages: 2 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 61 (Actual)
Dates: Start 2000-11; Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Bone Formation Rate | 8 months

SECONDARY OUTCOMES:
Bone histomorphometric parameters other than bone formation rate, biochemical parameters (phosphorus, calcium, PTH, alkaline phosphatase, FGF-23, vitamin D dose) | 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Isidro B Salusky, MD, Principal Investigator — University of California, Los Angeles

REFERENCES:
- [Derived] Natale P, Green SC, Ruospo M, Craig JC, Vecchio M, Elder GJ, Strippoli GF. Phosphate binders for preventing and treating chronic kidney disease-mineral and bone disorder (CKD-MBD). Cochrane Database Syst Rev. 2025 Jun 27;6(6):CD006023. doi: 10.1002/14651858.CD006023.pub4. PMID 40576086